CLINICAL TRIAL: NCT03597451
Title: The Effects of Extremity and "Core" Muscles Strength on Walking and Sit-to-Stand Performance in Patients With Multiple Sclerosis
Brief Title: The Effects of Muscles Strength on Physical Performance in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Principal Investigator, Gazi University
Other Study IDs: 435
Record Dates: First submitted 2018-07-09; First posted 2018-07-24 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
Keywords: strength; walking; sit-to-stand
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple sclerosis: Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS)
- Control: Healthy individuals of similar age and sex to patients

SUMMARY:
Muscle weakness, which is one of the most common symptoms in patients with MS, limits the activities of daily life activities of patients by causing balance and gait disturbance. Lower extremity muscle strengths of MS patients are reported to be weaker than healthy individuals. Broekmans et al. showed that the weakness of the knee flexor and extensor muscles in patients with MS caused a decrease in walking distance and they are important determinants of walking capacity.

The effects of the endurance and strength of core muscles, as well as the extremity muscles, are important on physical performance. The weakness of the extremities and core muscles in MS patients also affects the sit-to-stand performance negatively as well as a decrease in walking speed and capacity.

In this study, it was aimed to investigate the effects of extremity and core muscle strength on walking and sitting-up performance of MS patients.

DETAILED DESCRIPTION:
Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS) and healthy individuals of similar age and sex to patients will be included in the study. The strength of the extremity and core muscles, walking capacity, and sit-to-stand performance will be evaluated once.

Investigators will use descriptive statistics and t-tests to compare variables between groups. Investigators will examine the correlations between variables using Pearson bivariate correlations. The significance level is set at p<0,05

ELIGIBILITY:
Inclusion Criteria:

* Participants who 18-65 years of age
* MS patients who are ambulatory (Expanded Disability Status Scale score ≤ 5,5 ) in a stable phase of the disease, without relapses in the last 3 month.

Exclusion Criteria:

* Participants who have orthopedic, vision, hearing, or perception problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS patients who are ambulatory
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
strength of extremity muscles | baseline
  The isometric strength of lower extremity muscles will be assessed respectively using a hand-held dynamometer (Baseline®, White Plains, New York, USA).

SECONDARY OUTCOMES:
6 minutes walking test | baseline
  The Six-Minute Walking Test (6MWT) was performed to determine walking capacity.
timed up and go test | baseline
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
sit-to-stand test | baseline
  In this test, the participants will stand up from and sit down on 43 cm high armless chair as quickly as possible 5 times.
Side Bridge Test (core muscles endurance) | baseline
  The subjects were asked to lay on their left or right sides and to extend their legs fully. Then The subjects are asked to create a straight line with their body by lifting their hip from the floor.The measurements are recorded with a chronometer as seconds. The tests end when the subjects break the test positions.
Modified Biering-Sorensen test (core muscles endurance) | baseline
  In this test, the subjects are asked to lie down on a workout bench, aligning their anterior superior iliac spine with the edge of the bench, which allowed the upper body to be planked out over the edge. The subjects are asked to fold their arms on their chest and to put their hands on their shoulders. The measurements are recorded with a chronometer as seconds. The tests end when the subjects break the test positions.
Trunk Flexion Test (core muscles endurance) | baseline
  This test is initiated when the subjects are in a sit-up position with their back resting against a wedge that was angled 55° from the floor. The measurements are recorded with a chronometer as seconds. The tests end when the subjects break the test positions.
Prone bridge test (core muscles endurance) | baseline
  In this test, the subjects put their elbows on the ground as the starting position and open their feet about the width of their hips while keeping their body straight as they are required not to arch or bow. The measurements are recorded with a chronometer as seconds. The tests end when the subjects break the test positions.

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yahia A, Ghroubi S, Mhiri C, Elleuch MH. Relationship between muscular strength, gait and postural parameters in multiple sclerosis. Ann Phys Rehabil Med. 2011 May;54(3):144-55. doi: 10.1016/j.rehab.2011.02.004. Epub 2011 Mar 9. English, French. PMID 21493176
- [Background] Broekmans T, Gijbels D, Eijnde BO, Alders G, Lamers I, Roelants M, Feys P. The relationship between upper leg muscle strength and walking capacity in persons with multiple sclerosis. Mult Scler. 2013 Jan;19(1):112-9. doi: 10.1177/1352458512444497. Epub 2012 May 4. PMID 22562952
- [Background] Ketelhut NB, Kindred JH, Manago MM, Hebert JR, Rudroff T. Core muscle characteristics during walking of patients with multiple sclerosis. J Rehabil Res Dev. 2015;52(6):713-24. doi: 10.1682/JRRD.2015.01.0006. PMID 26562753
- [Background] Fry DK, Huang M, Rodda BJ. Core muscle strength and endurance measures in ambulatory persons with multiple sclerosis: validity and reliability. Int J Rehabil Res. 2015 Sep;38(3):206-12. doi: 10.1097/MRR.0000000000000109. PMID 25647356
- [Background] Bliss LS, Teeple P. Core stability: the centerpiece of any training program. Curr Sports Med Rep. 2005 Jun;4(3):179-83. doi: 10.1007/s11932-005-0064-y. PMID 15907272